CLINICAL TRIAL: NCT05004415
Title: An Open-Label, Single-Dose Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of [14C]-AT-527 in Healthy Adult Male Subjects
Brief Title: Mass Balance Study of AT-527 in Healthy Adult Male Subjects (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-006
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Intervention Model Description: Open-Label, Single-Dose pharmacokinetic (PK) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AT-527 550 mg (R07496998) (Experimental)
  Interventions: Drug: AT-527 (R07496998)

INTERVENTIONS:
Drug: AT-527 (R07496998) — Study participants will receive a single radiolabeled dose of 550 mg AT-527.

SUMMARY:
Mass balance study of AT-527 in Healthy Male Subjects.

DETAILED DESCRIPTION:
This is an open-label, single-dose study assessing the absorption, metabolism, excretion, and mass balance of [14C]-AT-527 in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/m2
* No clinically significant diseases captured in the medical history or clinically significant findings at screening physical examination.
* A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to dosing. A male who has been vasectomized less than 4 months prior to dosing must follow the same restrictions as a non-vasectomized male).
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy, adult male, 19-55 years of age, inclusive, at the screening visit.
Enrollment: 6 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Mass Balance | Day 1 to Day 15
  Total radioactivity recovery in urine and feces
Mass Balance | Day 1 to Day 15
  Percent of radioactive dose excreted in urine and feces

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Lincoln, Nebraska, United States